CLINICAL TRIAL: NCT02825524
Title: Efficacy and Safety of Endobiliairy Radiofrequency (Probe Habib TM EndoHPB) for the Destruction of Residual Endo Biliairy Dysplastic Buds After Endoscopic Ampullectomy: Prospective Multicenter Study
Brief Title: Destruction of Residual Endo-biliary Dysplastic Buds After Endoscopic Ampullectomy
Acronym: endoHPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Cochin (Other)
Responsible Party: Principal Investigator, Frederic PRAT, clinical professor, Hôpital Cochin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-A00721-40
Record Dates: First submitted 2016-06-15; First posted 2016-07-07 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Adenoma, Bile Duct
MeSH Terms: conditions — Adenoma, Bile Duct

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endobiliary radiofrequency (Experimental)
  Interventions: Device: Habib™ EndoHBP

INTERVENTIONS:
Device: Habib™ EndoHBP — During an endoscopic retrograde cholangiography, endobiliary application of radiofrequency through a dedicated probe named Habib.

SUMMARY:
The purpose of the study is to assess the efficacy and morbidity of biliairy radiofrequency ablation for the treatment of dysplastic endobiliairy residual lesions (low-grade dysplasia or high-grade dysplasia) after endoscopic ampullectomy for ampullary adenoma.

DETAILED DESCRIPTION:
Neoplastic lesions may persist at the termination of the common bile duct or pancreatic duct, after endoscopic ampullectomy for adenoma. Such lesions conduct to a difficult therapeutic problem because surgery (pancreaticoduodenectomy or trans-duodenal resection) has significant morbidity compared to non-invasive lesions. The use of endoscopic destruction techniques of dysplastic lesions, including radio-frequency could be an interesting alternative to reduce the risk of invasive cancer with less morbidity. Ablation with radio-frequency (RF) is a technique of local tissue destruction in use in many applications, percutaneously or intraoperatively for the treatment of hepatocellular carcinoma smaller and more recently for the endoscopic treatment of high-grade dysplasia of Barrett's esophagus. An RF probe has been developed for an endo-biliary application (Habib EndoHPB, Emcision) and 2 preliminary studies have reported the use in humans, in the indication of unresectable cholangiocarcinoma. These two studies have confirmed the feasibility of the technique, with few side effects and probable anti-tumor efficacy demonstrated by expanding the area of stenosis after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Presence of lesions of low-grade dysplasia (LGD) or high grade (HGD) in the common bile duct, confirmed by two pathological readings in relation to residual adenomatous tissue into the common bile duct after endoscopic ampullectomy for ampullome conducted in the previous year
* Lack of residual adenomatous lesion on the duodenal side after ampullectomy and possibly additional procedures (endoscopic mucosal resection or argon plasma). (excluding other duodenal adenomatous lesions in the context of familial adenomatous polyposis
* Consultative multidisciplinary digestive cancer meeting confirming the indication of treatment with endo-biliary radio-frequency
* Dysplastic lesions extending over 20 mm length maximum in the common bile duct
* Patients aged ≥ 18 years old and ≤ 85 years old
* Patients who consented to participate in the study
* No anesthesia contraindication (ASA 1,2,3)
* Patient affiliated to a social security scheme (beneficiary or legal)
* Lack of pregnancy and contraception being women age procreate

Exclusion Criteria:

* Lesions of invasive carcinoma in a patient whose clinical condition allows to consider a pancreaticoduodenectomy
* Endo-biliary dysplastic lesions diffuse or multifocal
* Presence of non extractable metal biliary expansive prosthesis
* History of pancreaticoduodenectomy or hepaticojejunostomy anastomosis
* Impassable stenosis of the common bile duct
* Severe coagulopathy, thrombocytopenia < 75,000 G/L , Clopidogrel treatment impossible to stop temporarily
* Anesthesia contraindication ( ASA 4)
* Pace maker or other active implantable medical device
* Inability to obtain informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-11; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
number of residual neoplasia | one year

SECONDARY OUTCOMES:
presence of low grade dysplasia or high grade dysplasia or invasive carcinoma | 6 months
number of surgery | one year
fever | 48 hours post endoscopic procedure
pain | 48 hours post endoscopic procedure
  Visual Analogue Scale
bleeding | 48 hours post endoscopic procedure
  hematemesis, hematochezia or melena or decreased more than 2 points of hemoglobin
acute pancreatitis | 48 hours post endoscopic procedure
  pain and increased of lipase more than 3 fold
cholangitis | 48 hours post endoscopic procedure
  fever and abnormal hepatic blood tests
perforation | 48 hours post endoscopic procedure
  pneumoperitoneum, retropneumoperitoneum, pneumothorax

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Camus M, Napoleon B, Vienne A, Le Rhun M, Leblanc S, Barret M, Chaussade S, Robin F, Kaddour N, Prat F. Efficacy and safety of endobiliary radiofrequency ablation for the eradication of residual neoplasia after endoscopic papillectomy: a multicenter prospective study. Gastrointest Endosc. 2018 Sep;88(3):511-518. doi: 10.1016/j.gie.2018.04.2332. Epub 2018 Apr 13. PMID 29660322